CLINICAL TRIAL: NCT04000243
Title: Interobserver Agreement of Endoscopic Diagnosis of Helicobacter Pylori Based on the Arrangement of Gastric Collecting Venules: Prospective and Multicenter Study
Brief Title: Diagnosis of Helicobacter Pylori Based on Gastric Collecting Venules
Status: Completed | Type: Observational
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Ana García-Rodríguez, Co-investigator (collaborator), Hospital Clinic of Barcelona
Other Study IDs: RAC-M
Record Dates: First submitted 2019-06-21; First posted 2019-06-27 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Helicobacter Pylori Infection; Upper Endoscopy; Regular Arrangement of Collecting Venules

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Diagnostic Test: Endoscopic diagnosis of Hp — Detection of a regular arrangement of collecting venules (RAC) pattern in the lesser gastric curvature

SUMMARY:
Helicobacter pylori (Hp) is the major cause of gastritis and gastritis-associated diseases. Detection of a regular arrangement of collecting venules (RAC) pattern in the lesser gastric curvature correlates with negative Hp status with a sensitivity and negative predictive value (NPV) higher than 90% in Asian countries.

In a recent study carried out in our hospital, it has been shown that the presence of RAC pattern in the lesser gastric curvature, evaluated with high definition endoscopy, can accurately identify patients without Hp.

The aim of this study is to confirm the validity of the endoscopic diagnosis of Hp infection in the West by means of the RAC pattern in a multicenter prospective study and to evaluate interobserver variability before establishing its applicability in clinical practice.

DETAILED DESCRIPTION:
We designed a prospective study including patients who will undergo upper gastrointestinal endoscopy from July 2019 to June 2020 at the Endoscopy Unit of Hospital Clinic of Barcelona.

The Ethics Committee of Hospital Clinic of Barcelona approved the study.

Upper gastrointestinal endoscopies will be performed with high definition endoscopes (Olympus, Germany) without magnification by three endoscopists. One of the endoscopists is considered as an expert with more than 20 years of experience and prior training in Japanese centers. All the examinations will be performed with sedation controlled by an anesthesiologist. After the routine examination of the esophagus, stomach, and duodenum, close observation will be carried out at the distal part of the lesser curvature and pictures will be taken. The Olympus system will be used for image storing and text reporting.

The presence of a regular or irregular arrangement of collecting venules will be evaluated in real time during gastric exploration in the lower part of the lesser curvature of the gastric body with good insufflation, close to the incisura angularis. If minute red points were visible regularly and homogenously, the finding will be scored as RAC positive (RAC+). If this finding was absent or there was a patchy distribution at the site of close observation, it will be defined as RAC negative (RAC-).

The following baseline characteristics will be collected: age, sex, antibiotics, proton-pump inhibitors, non-steroidal anti-inflammatory drugs (NSAIDs), antithrombotic or anticoagulant use in the last two weeks, history of Hp eradication and detection of significant endoscopic findings (erosive duodenitis, non-erosive duodenitis, duodenal ulcer, erosive gastritis, gastric ulcer and signs of atrophic gastritis or intestinal metaplasia).

Hp infection status will be determined by mucosal biopsies. We will perform 5 samples for histological study according to Sydney criteria (2 in antrum, 1 in incisura angularis and 2 in gastric body); or 2 biopsies (1 in antrum and 1 in gastric body) for histology and immunohistochemical study for Hp. Patients were classified as Hp positive if one of these two tests are positive.

For the histological study, samples will be fixed in formalin and stained with hematoxylin and eosin for the evaluation of gastritis and with Giemsa for Hp status. The immunohistochemical study will be carried out systematically in the case of a negative histological study for Hp. The pathologist has access to the endoscopic diagnosis but not to RAC status.

Statistical analysis

The quantitative variables will be described by the mean and the standard deviation, while the qualitative variables by proportion. The sensitivity, specificity, positive predictive value (PPV), NPV and accuracy of RAC for the diagnosis of uninfected Hp patients will be calculated. 95% confidence interval will be calculated by using standard formula. Comparisons will be done using Chi-square test for categorical variables and t test for continuous variables. In addition, a multivariate logistic regression analysis will be carried out to assess the existence of predictive factors of RAC and the odds ratio (OR) was calculated to indicate the associated risk. P <0 .05 will be considered statistically significant. All statistical analyses will be performed using the SPSS, version 23 (SPSS Inc., Chicago, USA).

ELIGIBILITY:
Inclusion Criteria:

- Patients older than 18 years who have an upper gastrointestinal endoscopy

Exclusion Criteria:

* Taking antibiotics in the last 4 weeks
* Presence of alimentary or hematic remains that prevent the correct visualization of the mucosa
* Bleeding from the upper gastrointestinal tract
* History of portal hypertensive gastropathy or lymphoma
* History of partial or total gastrectomy
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years who have an upper gastrointestinal endoscopy that do not meet the exclusion criteria
Sampling Method: Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Performance characteristics of a regular pattern of collecting venules (RAC) for the diagnosis of infection by Helicobacter pylori | one year
  Number of patients with RAC / no RAC and infection by Helicobacter pylori

SECONDARY OUTCOMES:
Interobserver variability for the diagnosis of RAC | one year
  Agreement among different endoscopists regarding the diagnosis of RAC in the pictures obtained and saved during the gastroscopies.
  The agreement will be evaluated by Cohen's kappa coefficient
Accuracy of RAC in patients treated with proton pump inhibitors | one year
  Number of cases with RAC / no RAC and infection by Helicobacter pylori in the subgroup of patients treated with proton pump inhibitors

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Fernandez-Esparrach, PhD, Study Director — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic of Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided